CLINICAL TRIAL: NCT07006012
Title: An Exploratory Clinical Study to Evaluate the Safety and Cytodynamic Characteristics of RGL-305 in Patients With Lymphoma
Brief Title: RGL-305+ Lymphoma + Exploratory Clinical Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Rong Tao, Chief Physician, Fudan University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGL-305-IIT-Lymphoma
Record Dates: First submitted 2025-05-02; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Lymphoma Patients With Complete Response (CR) or Partial Response (PR) After Standard Treatment Had a Positive Minimal Residual Lesion (MRD)
Keywords: Lymphoma; DLBCL
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In the RGL-305 low dose group, 3 to 6 subjects were planned to be enrolled in each dose (Experimental)
  Interventions: Drug: RGL-305
- In the RGL-305 high dose group, 3 to 6 subjects were planned to be enrolled in each dose group (Experimental)
  Interventions: Drug: RGL-305

INTERVENTIONS:
Drug: RGL-305 — RGL-305 is administered intravenously with a recommended rate of 3-5 mL /min. The interval after the first administration was 3 weeks, and then every 2 weeks was a cycle, each cycle was given d1, and up to 5 cycles of cell transfusion were received.

SUMMARY:
This study is an open, prospective, dose-increasing exploratory clinical trial. To evaluate the safety, cytodynamics and initial efficacy of RGL-305 in patients with lymphoma. All enrolled lymphoma patients were required to achieve CR or PR and MRD positive after standard treatment, PR patients were required to have a Deauville score of 4, and all patients would receive RGL-305 cell reinfusion therapy.

DETAILED DESCRIPTION:
This study adopted a "3+3" dose escalation design. RGL-305 preset two dose groups: low dose and high dose , and each dose group planned to enroll 3 to 6 subjects. The first patient in each group was set as a sentinel subject and observed for at least 48 hours. After evaluation by the investigators, it was found that no important adverse reactions occurred (such as CRS ≥ grade 3, aGVHD, anaphylaxis, etc.), and the other subjects at this dose level could be administered. The DLT observation period was set to 21 days after the subject received RGL-305 for the first time, during which the subject continued to receive the same dose level of RGL-305 for 1 cycle every 2 weeks (Q2W) and the first day of each cycle (D1), receiving a total of up to 5 cycles of cell transfusion. Treatment until the end of the cycle, disease recurrence or disease progression, intolerable toxicity, initiation of a new anti-tumor therapy, death (whichever occurs first)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate in the study and sign a written informed consent
2. Age 18-75 years old (including the boundary value), gender is not limited;
3. Patients with pathologically confirmed lymphoma who have previously received at least one standard treatment. After the last treatment, patients with Lugano 2014 lymphoma efficacy evaluation criteria were CR or PR, and MRD was positive. Patients with PR were required to have a Deauville score of 4.
4. Be willing to provide blood or tissue samples required for cytodynamic and biomarker detection before and after treatment;
5. ECOG score is 0 or 1;
6. Expected survival ≥3 months;
7. The function of vital organs meets the following criteria:

   1. Neutrophil absolute value (ANC) ≥1.0×109/L;
   2. Platelet count (PLT) ≥80×109/L;
   3. Hemoglobin (Hb) ≥90g/L;
   4. International standardized ratio (INR<1.5), activated partial thromboplastin time (APTT) ≤1.5×ULN;
   5. Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN);
   6. Total bilirubin (TBIL) ≤1.5×ULN;
   7. Serum creatinine (Scr) ≤1.5×ULN;
   8. Left ventricular ejection fraction (LVEF) ≥45%;
   9. Electrocardiogram: Fridericia corrected QT interval (QTcF) <470 ms; The QTc interval must be corrected according to Fridericia's standard with the correction formula QTcF=QT/RR^0.33.
8. Fertile female subjects must agree to effective contraception and refrain from egg donation for 6 months from the signing of the informed consent until the last administration of the investigational drug, the serum pregnancy test must be negative within 7 days prior to the first administration, and they are not lactating; Male subjects whose partner is a fertile woman must agree to highly effective contraception and refrain from sperm donation from signing the informed consent until 6 months after the final administration of the investigational drug (see Annex 6 for details)

Exclusion Criteria:

1. Previous adoptive cell therapy, including but not limited to tumor-infiltrating lymphocytes (TILs), chimeric antigen receptor T cells (CAR-T), and T cell receptor chimeric T cells (TCR-T);
2. Have previously received or planned to undergo organ transplantation or allogeneic stem cell or allogeneic bone marrow transplantation;
3. Combined with congenital or acquired immunodeficiency such as cellular immunodeficiency (e.g., DiGeorge syndrome, T-negative severe combined immunodeficiency [SSCID]) or combined T-cell and B-cell immunodeficiency (e.g., T-and B-negative combined immunodeficiency, Wiskott-Aldrich syndrome, ataxic telangiectasia, often) See variable immune deficiency); Or infected with human immunodeficiency virus (HIV);
4. The presence of autoimmune diseases, except for patients with hypothyroidism due to autoimmune thyroiditis who only need hormone replacement therapy;
5. History of epilepsy or other central nervous system diseases, or lymphoma invading the central nervous system;
6. Complicated with other malignant tumors, except malignant tumors with disease-free survival of more than 3 years and carcinoma in situ;
7. History of allergy to blood products, known to be allergic to test substances;
8. Any non-hematological toxicity associated with previous treatment does not return to ≤ grade 1, except for hair loss and peripheral neurotoxicity;
9. Those who had undergone major surgery (≥ Grade 3 surgery) within 4 weeks before the start of study treatment, or who required elective surgery during the trial period;
10. Have an poorly controlled or severe cardiovascular disease, such as symptomatic congestive heart failure (NYHA class III or IV), a myocardial infarction within 6 months prior to study initiation, or unstable angina within 1 month prior to study initiation, or an arrhythmia requiring treatment or intervention, Or hypertension remains poorly controlled after adequate treatment (systolic blood pressure ≥150mmHg, diastolic blood pressure ≥90mmHg);
11. Known hereditary or acquired bleeding or thrombotic tendencies;
12. Subjects with a known or highly suspected history of interstitial pneumonia, or evidence of active interstitial pneumonia on chest CT during the pre-screening period; Known history of idiopathic pulmonary fibrosis, institutional pneumonia (such as bronchiolitis obliterans or cryptogenic institutional pneumonia); Subjects who may interfere with the detection or management of suspected drug-related pulmonary toxicity;
13. A severe infection occurring within 28 days prior to study initiation (such as intravenous antibiotics, antifungal, or antiviral drugs as required by clinical practice), or an active infection receiving therapeutic intravenous or oral antibiotics within 14 days prior to study initiation, or an unexplained fever;
14. Active hepatitis B (HBV), hepatitis C (HCV), cytomegalovirus (CMV), EB virus (EBV), HIV, syphilis infection;
15. Plan to receive live attenuated vaccine (inactivated vaccine is allowed) within 28 days before the start of study treatment or during the study period and 90 days after the end of study drug treatment;
16. In the investigator's judgment, the subject has other factors that may affect the study results or lead to the forced termination of the study treatment;
17. During the study period, subjects considering fertility, female subjects became pregnant or breastfed within 6 months of the last study drug administration.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of RGL-305 | up to 2 years
  Incidence and severity of adverse events (AE)/serious adverse events (SAE) (severity based on CTCAE v 5.0 criteria) and association of adverse events with the investigational drug
  - Dose limiting toxicity (DLT) incidence of DLT during the observation period

SECONDARY OUTCOMES:
To evaluate the cytodynamics of RGL-305 after reinfusion | up to 2 years
  Flow cytometry was used to detect the number and proportion of Target cells in peripheral blood and the changes compared with baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rong Tao, M.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No